CLINICAL TRIAL: NCT04812275
Title: Absorbable or Non Absorbable Sutures in Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Hand surgery Södersjukhuset (Other)
Responsible Party: Principal Investigator, Mirjam Hägg, Resident Physician, Department of Hand surgery Södersjukhuset
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06004
Record Dates: First submitted 2021-02-26; First posted 2021-03-23 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Wound Complication Hand Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non absorbable suture (Active Comparator): Wound closure with non absorbale suture. Dimension and brand at the discretion of the surgeon.
  Interventions: Procedure: Skin closure
- Absorbable suture (Experimental): Wound closure with absorbale suture. Dimension and brand at the discretion of the surgeon.
  Interventions: Procedure: Skin closure

INTERVENTIONS:
Procedure: Skin closure — Skin closure

SUMMARY:
After all surgical procedures, the skin must be closed with some form of stitch, in healthcare called suture. According to the tradition of hand surgery, sutures that must be removed by caregivers, ie non-resorbable thread, have been used extensively, and the frequency of complications in the form of wound rupture and infection is low. For many procedures, however, it can be an advantage to avoid removing the stitches, as it is both painful for the patient and time-consuming and resource-consuming for both the patient and the healthcare system. You can then use a thread that the body itself breaks down and absorbs, ie resorbable suture. In the project, we will compare resorbable and non-resorbable suture with the primary outcome of superficial infection in the surgical area sometime day 1-20 after surgery. Secondary outcomes are the occurrence of wound rupture, pain VAS (Visual Analog Scale) when changing 2 weeks postoperatively, patient satisfaction VAS at 2 weeks and time spent in minutes for changing at 2 weeks postoperatively. The project will include all consecutive patients> 18 years of age who are operated on at the hand surgery clinic Södersjukhuset for elective or emergency surgery that do not meet the exclusion criteria. The project will include 270 patients.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients> 18 years of age who are operated on at the hand surgery clinic Södersjukhuset for elective or emergency surgery that do not meet any of the exclusion criteria.

Exclusion Criteria:

* -The researcher has an age <18 years.
* Patients with known healing problems in the past, for example patients with burns or during cortisone treatment.
* Patients undergoing surgery where skin grafting occurs.
* Patients with acute injuries that include a traumatic wound-ie what is usually referred to as "open injuries" -where the risk of infection is higher from the beginning.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Infection | 2 weeks
  Signs of superficial infection after surgery. Redness, pus, swelling.

SECONDARY OUTCOMES:
Rupture | 2 weeks
  The prevalens of wound rupture after hand surgery
VAS | 2 weeks
  Visual analog scale
Time | 2 weeks
  Time consumption removal of sutures

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No